CLINICAL TRIAL: NCT02799446
Title: Efficacy of Reslizumab for the Treatment of Chronic Rhinosinusitis A Double Blind, Randomized, Placebo-controlled, Phase III Trial
Brief Title: Effect of Reslizumab in Chronic Rhinosinusitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joshua S. Jacobs (Other)
Responsible Party: Sponsor-Investigator, Joshua S. Jacobs, MD, Allergy and Asthma Clinical Research Inc.
Organization: Allergy and Asthma Clinical Research Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AACR-01
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Sinusitis
Keywords: sinusitis, rhinitis, rhinosinusitis, chronic
MeSH Terms: conditions — Sinusitis; Rhinitis; Rhinosinusitis; Bronchiolitis Obliterans Syndrome | interventions — reslizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Reslizumab (Experimental): Reslizumab will be administered intravenously every 4 weeks at a dose of 3mg/kg.
  Interventions: Drug: Reslizumab
- Placebo (Placebo Comparator): Matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reslizumab — Reslizumab 3mg/kg intravenous (IV)
  Arms: Reslizumab
Drug: Placebo — Matching Placebo intravenous (IV)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Reslizumab is effective for the treatment of chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Willingness and ability to comply with the requirements of the study
3. Female or male patients ages 18-75 at the time of screening
4. A diagnosis of chronic rhinosinusitis according to the clinical practice guideline (update) of the American academy of otolaryngology - head and neck surgery
5. Elevated blood eosinophils
6. Significant findings on computed tomography (CT) scan

Exclusion Criteria:

1. Unable to sign informed consent form
2. A woman that is pregnant or nursing a child
3. Known hypersensitivity to Reslizumab
4. Active cigarette smoking in the year prior to screening
5. Known underlying immunodeficiency
6. History of alcohol or drug abuse in the year prior to screening

Other criteria may apply. Please contact the investigator for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in computed tomography (CT) score | 24 weeks

SECONDARY OUTCOMES:
Quality of life questionnaire | 24 weeks
Smell test | 24 weeks
Endoscopy score | 24 weeks
Adverse events by body system | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Jacobs, MD, Principal Investigator — Allergy and Asthma Clinical Research
Locations (1):
- Allergy and Asthma Clinical Research, Walnut Creek, California, United States